CLINICAL TRIAL: NCT07388446
Title: Role of Mucosal Associated Invariant T Cells in Hidradenitis Suppurativa
Brief Title: MAIT Cells in Hidradenitis Suppurativa
Acronym: HS-MAIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL25-0435; 2025-A01606-43 (Other: ID-RCB)
Record Dates: First submitted 2026-01-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis suppurativa; physiopathology; immunology; Mucosal Associated Invariant T cells
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hidradenitis suppurativa patients (Experimental): * Age 18 to 65 years
  * Ability to give informed consent and comply with protocol
  * Health insurance coverage
  * For women of childbearing potential: negative pregnancy test
  * Diagnosed for ≥ 6 months
  * IHS4 ≥ 4
  * Planned treatment with adalimumab, secukinumab, or bimekizumab within 7 days
  * Normal chest imaging and negative quantiferon and viral serologies (HIV, HBV, HCV) within 6 months
  * Presence of at least one active inflammatory lesion located outside a strict anatomical fold and outside the face, which will be preferentially selected for lesional skin biopsy.
  Interventions: Other: Collect lesional biopsies; Other: Collect score from Bristol stool scale
- Control patients (Active Comparator): * Age 18 to 65 years
  * Ability to give informed consent and comply with protocol
  * Health insurance coverage
  * For women of childbearing potential: negative pregnancy test
  * Diagnosis of plaque psoriasis or back-acne or impetigo
  Interventions: Other: Collect lesional biopsies; Other: Collect score from Bristol stool scale

INTERVENTIONS:
Other: Collect lesional biopsies — For HS and control patients (psoriasis, acne, impetigo): perform two skin biopsies :
  * a 6-mm skin biopsy on a lesional area (lesion, V1)
  * a 6-mm skin biopsy on a non-lesional area (non-lesional, V1) Lesional biopsies will be performed on lesions located outside a strict anatomical fold and outside the face, in accordance with regulatory requirements for category 2 research.
Other: Collect score from Bristol stool scale — Collect score from Bristol stool scale and give stool collection kit to all patient

SUMMARY:
Hidradenitis Suppurativa (HS) is a chronic, debilitating inflammatory skin disease characterized by painful, purulent lesions primarily in skin folds. Its pathogenesis remains poorly understood. The clinical benefit observed with both antibiotics and immunosuppressive therapies suggests HS may involve an abnormal immune response to skin microbiota.

Mucosal-associated invariant T (MAIT) cells are immune cells that bridge innate and adaptive immunity and are known to regulate microbial flora. Dysfunctional MAIT cells have been implicated in autoimmune diseases such as type 1 diabetes, inflammatory bowel diseases, and psoriasis. Preliminary data from the VERIMMUNE study (NCT05735925) indicate that HS patients show a depletion of circulating MAIT cells and increased infiltration of CD8+ MAIT cells in lesions, associated with reduced activation and greater disease severity. These findings support the hypothesis that MAIT cell dysfunction plays a central role in HS and may serve as a biomarker for treatment response. This exploratory study aims to (Primary) characterize the phenotype and frequency of MAIT cell subsets in the skin and blood of HS patients compared to controls with other inflammatory skin diseases (psoriasis and back-acne); and to determine whether MAIT cell phenotype before treatment predicts clinical response to biologic agents.

The study will recruit adults (18-65 years) with moderate-to-severe HS and matched controls with plaque psoriasis, or back-acne, or impetigo. All HS participants must be biologic-naïve at baseline and will be treated per national guidelines (adalimumab, secukinumab, or bimekizumab). No therapeutic intervention is imposed; patients are followed according to usual care. Skin and blood samples will be collected before and after treatment to assess immune profiles.

To minimize bias HS patients will be age/sex-matched with controls; only patients with active, inflammatory HS lesions will be included; controls were selected to represent related yet distinct pathologies: back-acne (follicular but distinct mechanism), psoriasis (different lesion type, shared type-17 inflammation) and impetigo (skin bacterial infection).

The Immunophenotyping strategy will use high-dimensional flow cytometry (Cytek® Aurora); researchers will analyze immune cell subsets (e.g., B cells, γδ T cells, NK cells, ILCs, MAIT, NK-T) in skin and blood. Specific markers for activation (CD69, PD-1, ICOS), differentiation (CCR7, CD45RA), proliferation (Ki-67), cytokine receptors, and chemokines will be assessed.

The primary endpoint will be the frequency of MAIT cells in lesional vs. non-lesional skin and blood compared to controls before and after 12 weeks of biologic agent. The secondary endpoints will be changes in MAIT cell phenotype after 12 weeks of treatment, correlation with clinical improvement (defined by IHS4-55 response: ≥55% reduction in IHS4 score) and MAIT cell functions (assessed in vitro before and after treatment, anti-bacterial activity, capacity to proliferate and to be activated).

This is a prospective, monocentric, exploratory study with intra-individual comparison and external active controls. The study falls under category 2 (interventional research with minimal risks). Clinical data, biopsy samples, and immune profiles will be collected before and after biologic therapy in moderate-to-severe HS patients (IHS4 ≥4), biologic-naïve, eligible for biologic agents treatment, with no antibiotics or immunosuppressive drugs in the prior month. The controls will be adults with psoriasis or back-acne or impetigo (no follow-up for control patients).

This study has no direct therapeutic benefit for participants. However, it offers detailed clinical follow-up and may significantly improve understanding of HS pathogenesis. Known procedural risks (local anesthesia, biopsy, venipuncture) are minimal and mitigated through standard precautions and inclusion criteria.

Expected benefits and impact : clarify the role of MAIT cells in HS pathophysiology; identify novel immune biomarkers predictive of biologic therapy response; support future therapeutic stratification and personalized treatment approaches in HS.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 to 65 years (included)
* Subject able to read, understand and give documented informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subject with health insurance coverage according to local regulations
* For woman with childbearing potential, negative pregnancy test at the inclusion visit Specific criteria for HS patients
* Subject diagnosed with HS for at least 6 months
* Subject diagnosed with moderate-to-severe HS defined by IHS4 score > 4
* Subject is planned to be treated within 7 days with either adalimumab or secukinumab or bimekizumab under the conditions defined by the French National Health Authority
* Normal chest imaging within 6 months prior to inclusion.
* Negative Quantiferon test within 6 months prior to inclusion.
* Negative HIV, HBV, and HCV serologies within 6 months prior to inclusion.
* Presence of at least one active inflammatory lesion located outside a strict anatomical fold and outside the face, which will be selected for lesional skin biopsy Specific criteria for control patients
* Subject diagnosed with plaque psoriasis or back-acne or impetigo

Exclusion Criteria:

* - Pregnancy or breast-feeding women
* Subject treated by immunosuppressive/immunomodulatory substances including oral corticosteroid or biological agents within 4 weeks before inclusion
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the assessment or put the subject at risk
* Linguistic or mentally incapacity to sign the consent form
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial
* Weight <50 kg
* Diabetes
* Specific treatments such as metformin or GLP1-agonist that may interfere with MAIT cell activity
* History of allergic reaction to local anesthetic product
* History of wound healing disorders (e.g. hypertrophic scars, keloids)
* Subject treated by oral or topical antibiotics within 2 weeks before inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of MAIT cells within CD45+ cells in the blood of HS patients | Before and after 12 weeks initiating biotherapy treatment of HS patients.
  Frequency of MAIT cells within CD45+ cells in the blood of HS patients before and after treatment

SECONDARY OUTCOMES:
Frequency of MAIT cells in skin and blood of HS patients | Before and after 12 weeks of biotherapty treatment of HS patients
  Frequency of MAIT cells in skin and blood HS patients comparing lesional and non lesional skin
Phenotype of MAIT cells in skin and blood | Before and after 12 weeks of biotherapty treatment of HS patients
  Level of expression of activation markers of MAIT cells such as CD69
Characterize antibacterial activity of MAIT cells in the skin and blood | Before and after 12 weeks of biotherapty treatment of HS patients
  MAIT cells will be isolated from skin and peripheral blood and co-cultured with MR1⁺ HeLa cells or primary keratinocytes previously infected with E. coli. Antibacterial activity will be assessed by quantifying viable bacteria using colony-forming unit (CFU) assays, with antibacterial activity expressed as the percentage and log₁₀ reduction of viable bacteria relative to control conditions without MAIT cells.
Proliferation capacity of MAIT cells | Before and after 12 weeks of biotherapy treatment of HS patients
  Expression of Ki67 in vitro after stimulation
Charaterize microbial composition in stool | Before and after 12 weeks of biotherapy treatment of HS patients
  Level of expression of activation markers of MAIT cells

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Dermatologie - CLIMA Pav R, Lyon, France